CLINICAL TRIAL: NCT04585061
Title: A Novel Approach in Reducing Dental Pain and Anxiety of Pediatric Patient During Local Anesthesia. A Clinical Experimental Study
Brief Title: A Novel Approach in Reducing Dental Pain and Anxiety of Pediatric Patient During Local Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Abdulrahman Alasmari, Principal Investigator, Riyadh Elm University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FPGRP/2020/489/269
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Lidocaine; Xylitol

STUDY DESIGN:
Intervention Model Description: Randomized Intervention Model: Split-mouth assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sweet test group (Active Comparator): Local anesthesia with conventional syringe Procedure: Local anesthesia with conventional syringe + xylitol sublingual tablet Buccal infiltration in posterior maxillary region with traditional technique. A 27 gauge short needle is inserted in the mucobuccal fold above the tooth to be anesthetized.
  Interventions: Drug: Lidocaine Hydrochloride; Dietary Supplement: Xylitol
- Virtual reality group (Active Comparator): Local anesthesia with conventional syringe + VR device Device: Local anesthesia with conventional syringe + VR device Virtual reality device (Harga Miniso Vr Glass 3d terbaru) is placed on the face of the patient, playing a video of Tom and Jerry cartoon.
  Buccal infiltration in posterior maxillary region with traditional technique. A 27 gauge short needle is inserted in the mucobuccal fold above the tooth to be anesthetized.
  Interventions: Drug: Lidocaine Hydrochloride; Device: Virtual reality device (Harga Miniso Vr Glass 3d terbaru)

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — 1.8ml of 2%Lidocaine HCl to be administered via a 21mm needle
  Other Names: lignocaine
Device: Virtual reality device (Harga Miniso Vr Glass 3d terbaru) — Virtual reality device (Harga Miniso Vr Glass 3d terbaru) is placed on the face of the patient, playing a video of Tom and Jerry cartoon.
  Buccal infiltration in posterior maxillary region with traditional technique. A 27 gauge short needle is inserted in the mucobuccal fold above the tooth to be anesthetized
  Other Names: VR
  Arms: Virtual reality group
Dietary Supplement: Xylitol — Buccal infiltration in posterior maxillary region with traditional technique. A 27 gauge short needle is inserted in the mucobuccal fold above the tooth to be anesthetized while xylitol tablet putted under tongue
  Other Names: Xylitol candy
  Arms: sweet test group

SUMMARY:
The aim of this study is to determine the efficacy of sweet in compare to virtual reality (VR) device in reducing injection pain and anxiety associated with local anesthesia in pediatric dental patients.

The clinical trial is a randomized split-mouth assignment. Included patients are 5 - 12 years old requiring local anesthetic infiltration with conventional syringe (CS) for conservative treatment of two primary maxillary molars bilaterally.

Eligible patients undergo two single-visit treatments after CFSS-DS measurement before each, whereas sweet is allocated to first local anesthesia procedure and VR is allocated to second local anesthesia procedure. Primary outcome measure will be pain felt during injection, reported by patient on visual analogue scale (VAS). Secondary outcome measures: self-reported anxiety during injection on FIS; pain-related behavior according to FLACC scale; heart-rate dynamics; patient preference to local anesthesia method - CS+sweet or CS+VR.

DETAILED DESCRIPTION:
Achieving local anesthesia in children is one of the critical aspects of pain management and they effect the quality of treatment as well as behavior of child.

A contemporary engaging form of distraction is represented by virtual reality devices. Virtual reality (VR) devices create a virtual environment of view and sound that allow patients to be immersed in an interactive, simulated world to distract them from pain. The VR devices have a wide viewing field and three-dimensional displays that project the images right in front of the user. They not only show potentially attractive audio-visual stimuli, but also exclude all other visual environmental stimuli that may affect the patient.

While sweet-tasting reduce signs of pain during painful procedures. This effect is considered to be mediated both by the release of endorphins and by a pre absorptive mechanism related to the sweet taste.

The aim of this study is to determine the efficacy of sweet-testing compare to a virtual reality (VR) device in reducing injection pain and anxiety associated with local anesthesia in pediatric dental patients.

The device used in this study is Harga Miniso Vr Glass 3d terbaru, compatible with a mobile phone.

The sweet used is xylitol tablet The clinical trial is a randomized split-mouth assignment. Included patients are healthy positive children 5-12 years old requiring local anesthetic infiltration for conservative treatment of two primary maxillary molars bilaterally.

Eligible patients undergo two single-visit treatments after measurement of dental fear prior to each according to the Dental Subscale of the Children's Fear Survey Schedule (CFSS-DS). Local anesthetic is delivered through buccal infiltration with conventional syringe, where is the sweet-test applied with first local anesthesia procedure and the virtual reality distraction is allocated to second local anesthesia procedure. Primary outcome measure will be pain felt during injection, reported by patient on visual analogue scale. Secondary outcome measures: self-reported anxiety during injection on Facial Image Scale; pain-related behavior according to Faces, Legs, Activity, Cry, Consolability (FLACC) scale; heart-rate dynamics; patient preference to local anesthesia method - sweet test infiltration or virtual reality device-assisted injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients, identified as positive or definitely positive through Frankl behavioral rating scale.
* Children, requiring local anesthesia infiltration for conservative treatment of two primary upper jaw molars bilaterally.
* Children without previous experience with local anesthesia for dental treatment.
* Obtained informed consent from parents or gave-givers to participate in the study.

Exclusion Criteria:

* Children who are considered medically compromised or medically complex patients. The absence of disease is confirmed by anamnestic interview with a parent or a care-giver of the child and excludes general acute or chronic disease, cognitive impairment, psychogenic non-epileptic events, sensitivity to flashing light or motion.
* Vision requiring correction with eyeglasses.
* Recent injury to the eyes or face that prevents comfortable use of VR hardware or software.
* Patients who are undergoing therapy with neurological, sedative, analgesic and/or anti-inflammatory drugs 7 days prior to treatment.
* Patients with allergy to local anesthetics, xylitol.
* Children, who are first time ever dental patients.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Pain felt during injection using visual analogue scale | Immediately after local anesthetic delivery
  Self-reported pain by the patient immediately after local anaesthesia infiltration using a VAS (visual analogue scale), containing a combination of Numeric Rating Scale (0-10, where 0 means no pain, 10 - worst possible pain) and Wong-Baker Faces Pain Scale, including pictures of facial expressions with correlating numbers of 0-10 (0 being 'no hurt' and 10 being 'hurts worst'). The combination allows children to pick a facial expression, that corresponds with their pain and see a number that matches it.

SECONDARY OUTCOMES:
Pain-related behavior evaluated on the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale | During local anesthesia procedure
  Evaluated by the outcomes assessor. The FLACC scale has five criteria - Faces, Legs, Activity, Cry, Consolability, which are each assigned a score of 0, 1 or 2. Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain
Self-reported anxiety during injection evaluated on FIS | Immediately after local anesthetic delivery
  The Facial Image Scale (FIS) comprises a row of five faces from very unhappy (score 5) to very happy (score 1).
Heart rate dynamics of the patient | Baseline (Start: in the waiting room), at least 5 minutes before local anaesthesia procedure. End: at least 5 minutes after treatment.
  Patient's left index finger is connected to a portable recording pulse oximeter for children.
Assessment of self-reported dental fear on CFSS-DS questionnaire | At least 5 minutes before local anesthesia
  After each procedure

CONTACTS AND LOCATIONS:
Overall Officials: AbdulRahman Alasmari, Resident, Principal Investigator — Riyadh Elm University
Locations (1):
- AbdulRahman Alasmari, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buchanan H, Niven N. Validation of a Facial Image Scale to assess child dental anxiety. Int J Paediatr Dent. 2002 Jan;12(1):47-52. PMID 11853248
- [Result] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Result] von Baeyer CL, Spagrud LJ. Systematic review of observational (behavioral) measures of pain for children and adolescents aged 3 to 18 years. Pain. 2007 Jan;127(1-2):140-50. doi: 10.1016/j.pain.2006.08.014. Epub 2006 Sep 25. PMID 16996689
- [Result] Malviya S, Voepel-Lewis T, Burke C, Merkel S, Tait AR. The revised FLACC observational pain tool: improved reliability and validity for pain assessment in children with cognitive impairment. Paediatr Anaesth. 2006 Mar;16(3):258-65. doi: 10.1111/j.1460-9592.2005.01773.x. PMID 16490089
- [Result] ten Berge M, Veerkamp JS, Hoogstraten J, Prins PJ. Childhood dental fear in the Netherlands: prevalence and normative data. Community Dent Oral Epidemiol. 2002 Apr;30(2):101-7. doi: 10.1034/j.1600-0528.2002.300203.x. PMID 12000350
- [Result] Keefe FJ, Rumble ME, Scipio CD, Giordano LA, Perri LM. Psychological aspects of persistent pain: current state of the science. J Pain. 2004 May;5(4):195-211. doi: 10.1016/j.jpain.2004.02.576. PMID 15162342
- [Result] Locker D, Thomson WM, Poulton R. Psychological disorder, conditioning experiences, and the onset of dental anxiety in early adulthood. J Dent Res. 2001 Jun;80(6):1588-92. doi: 10.1177/00220345010800062201. PMID 11499519
- [Result] Thomson WM, Locker D, Poulton R. Incidence of dental anxiety in young adults in relation to dental treatment experience. Community Dent Oral Epidemiol. 2000 Aug;28(4):289-94. doi: 10.1034/j.1600-0528.2000.280407.x. PMID 10901408
- [Result] Bikmoradi A, Khaleghverdi M, Seddighi I, Moradkhani S, Soltanian A, Cheraghi F. Effect of inhalation aromatherapy with lavender essence on pain associated with intravenous catheter insertion in preschool children: A quasi-experimental study. Complement Ther Clin Pract. 2017 Aug;28:85-91. doi: 10.1016/j.ctcp.2017.05.008. Epub 2017 May 24. PMID 28779942
- [Result] Zhang C, Qin D, Shen L, Ji P, Wang J. Does audiovisual distraction reduce dental anxiety in children under local anesthesia? A systematic review and meta-analysis. Oral Dis. 2019 Mar;25(2):416-424. doi: 10.1111/odi.12849. Epub 2018 Sep 21. PMID 29498793
- [Result] Messieha Z. Risks of general anesthesia for the special needs dental patient. Spec Care Dentist. 2009 Jan-Feb;29(1):21-5; quiz 67-8. doi: 10.1111/j.1754-4505.2008.00058.x. PMID 19152564